CLINICAL TRIAL: NCT02078570
Title: Breast Cancer Biomarker Sample Collection for the dtectDx v2 Assay Proof of Concept Protocol
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Provista Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: dtectDx-Breast-002
Record Dates: First submitted 2014-02-28; First posted 2014-03-05 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 35mL or 2 1/2 tablespoons of blood will be drawn from your arm

GROUPS / COHORTS (1):
- Breast Cancer ACR BI-RAD Category 3 or 4 result

SUMMARY:
The major purpose of this study is to evaluate a laboratory developed test that measures multiple breast cancer-specific biomarker proteins and multiple antibodies in your blood samples. The biomarker and antibody results along with your personal medical profile will be evaluated to determine your risk for the presence of a malignancy in the breast as compared to your breast evaluation assessment conducted by your physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult women from 25 years of age to below 75 years of age
* Breast evaluation results of ACR BI-RADS® Category 3 or 4 by imaging and physicians clinical and radiological evaluation
* Study visit and blood collection within 4 weeks (28 days) of ACR BI-RADS assessment
* Patient agrees to with additional health data being gathered at 6 months post assessment for diagnostic follow-up
* Samples collected under IRB approval and Informed Consent
* Testing performed under IRB approval or waiver (as applicable)
* Previous approved procedures to enroll patients: breast augmentation & cyst aspiration

Exclusion Criteria:

* Adults from 76 years of age or older and below 25 years of age
* Final breast evaluation results other than a ACR BI-RADS Category 3 or 4
* Subjects that have had a breast biopsy performed during the 6 months prior to the study visit
* Samples not collected under IRB approval and Informed Consent
* Testing not performed under IRB approval or waiver (as applicable)
* Prior breast cancer diagnosis.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinics
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Quantitative Protein Algorithmic Score (QPAS) | Baseline
  Part I: Establish an acceptable algorithm for the generation of a single numerical score from the combination of the 10 cancer biomarkers that comprise the dtectDx Breast v2.0 Assay Part II: Define a numerical score cutoff that differentiates malignant from nonmalignant breast cancer in this population of woman
Modified Quantitative Protein Algorithmic Score (QPAS) | 6 Months
  Demonstrate proof-of-concept for use of the dtectDx-Breast Assay to assess likelihood of breast cancer malignancy in conjunction with the physicians clinical and radiological evaluations.

SECONDARY OUTCOMES:
QPAS relative to BI-RADS | Baseline
  Demonstrate the numerical score, collaborated via proprietary algorithm , for the dtectDx-Breast Assay v2.0 increases the likelihood of malignant breast cancer detection when used adjunctively with the assessment of BI-RADS Categories 3 and 4 compared to the assessment of BI-RADS Categories 3 and 4 alone.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Sutter Institute, Sacramento, California
  - Scripps, San Diego, California
  - Henry Ford Hospital, Detroit, Michigan
  - Sinai Grace, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Summit Medical Group Breast Center New Jersey, Berkeley Heights, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Mercy Womens Center, Oklahoma City, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Avera Research Institute, Sioux Falls, South Dakota

REFERENCES:
- See also: Related Info — http://www.provistadx.com